CLINICAL TRIAL: NCT05176626
Title: Long-term Effectiveness of the Antiobesity Medication Phentermine
Acronym: LEAP
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Johns Hopkins University (Other); Kaiser Permanente (Other); HealthPartners Institute (Other); The University of Texas Health Science Center, Houston (Other); Biomedical Research Institute of New Mexico (Other); WW International Inc (Industry); KVK-Tech, Inc. (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00079100; UG3HL155801 (NIH)
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Obesity; Drug; Lifestyle, Healthy
Keywords: weight-loss; lifestyle intervention; phentermine
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Phentermine

STUDY DESIGN:
Intervention Model Description: Blinded, placebo-matched
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, study investigators and research staff, care providers, laboratory staff, and outcomes assessors will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phentermine (Experimental): Participants randomized to active treatment in LEAP will be provided with phentermine hydrochloride 8 mg scored tablets. This formulation of the drug is commercially available and marketed as Lomaira TM.
  Interventions: Behavioral: Online Lifestyle Behavioral Therapy; Drug: Phentermine Hydrochloride 8 MG
- Placebo (Placebo Comparator): Participants randomized to the control arm of LEAP will be provided with placebo tablets consisting of cellulose and corn starch and manufactured to have the same characteristics of the active drug, including size, shape, weight, and sensory perceptions.
  Interventions: Behavioral: Online Lifestyle Behavioral Therapy

INTERVENTIONS:
Behavioral: Online Lifestyle Behavioral Therapy — Participants will receive access to the WW™ digital application for the duration of their participation. The WW™ digital application can be accessed using a smartphone, tablet or personal computer and includes functions such as food journaling, progress charts, lifestyle coaching , ability to manually enter exercise data or link with a fitness tracking device, incentives for behavior change, recipes, and local restaurant recommendations using GPS. Over the course of 12 clinic visits with an obesity provider, participants will be prescribed a dietary plan based on the WW™ app and will be asked to journal dietary intake.
Drug: Phentermine Hydrochloride 8 MG — At the randomization visit, participants will be started on 8 mg PO daily of phentermine or placebo, with a recommendation to take the medication in the morning. They will be provided with detailed instructions on how to increase their dose of study drug over the subsequent weeks. After one week, participants will increase to 16 mg daily. After the second week, participants will further increase their dose to 24 mg daily and at the 1-month in-person follow-up, participants who tolerate the 24 mg dose will be maintained on this as the maximum daily dose for a total of 24 months. For participants who do not tolerate an escalation in medication dose due to side effects, adverse events, and/or elevations in blood pressure and/or heart rate, the study clinician may adjust the dose and/or delay dose escalation. Study clinicians will work with participants to achieve and sustain the maximum dose tolerated.
  Other Names: Lomaira
  Arms: Phentermine

SUMMARY:
The purpose of this research study is to understand the long-term effects of the drug phentermine on weight, blood pressure, other health outcomes, and safety. Phentermine has been approved by the US Food and Drug Administration (FDA) for weight management since 1959, but it has not been approved for long-term use (i.e., treatment lasting more than 12 weeks). This trial is designed to learn about the long-term effects of phentermine for up to 2 years because obesity is a chronic disease and expert guidelines recommend long-term use of anti-obesity medications as one treatment option.

DETAILED DESCRIPTION:
The Long-term Effectiveness of the Anti-obesity medication Phentermine (LEAP) trial, a placebo-controlled, randomized trial, will be conducted at 5 clinical sites across the United States. All participants will be provided with an evidence-based online lifestyle intervention, and participants receiving 24 mg/day of phentermine vs. a placebo for up to 24 months will be compared in an intent-to-treat fashion. The co-primary outcomes of percent weight loss and change in systolic blood pressure at 24 months will be examined. Also, between group changes in drivers of energy balance, including resting metabolic rate, caloric intake, physical activity and dietary composition will be compared. To explore the effects of weight loss on cardiometabolic health, changes in heart rate, hemoglobin A1c, lipids, waist circumference, atherosclerotic cardiovascular disease (ASCVD) risk score, and novel ECG markers of cardiac strain will be compared. Overall adverse event and serious adverse event rate, including rates of incident cardiovascular disease or death, will be measured.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-44.9 kg/m2 or BMI 27-29.9 with weight related comorbidity (including hypertension, prediabetes, type 2 diabetes mellitus, dyslipidemia, nonalcoholic fatty liver disease, treated obstructive sleep apnea, osteoarthritis, low back pain, gastroesophageal reflux disease)
* English-speaking
* Has a smartphone or other device with regular internet access
* Interested in and willing to lose weight as a result of treatment
* Able to take oral medication and willing to adhere to the clinical visit schedule for the trial and lifestyle based treatment regimen throughout the study duration, as recommended by the study clinician
* For females of reproductive potential: use of effective contraception for at least 1 month prior to randomization and agreement to use such a method during study participation and for an additional 8 weeks after the end of study drug administration
* Provision of electronically-signed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* History of coronary artery, cerebrovascular or peripheral arterial disease including myocardial infarction, unstable angina, revascularization, stroke/TIA, carotid intervention, claudication
* Poorly-controlled blood pressure (>149/94) or elevated heart rate (>110 bpm)
* History of cardiac arrhythmia
* Active / currently-treated hyperthyroidism
* History of glaucoma or been told by an ophthalmologist that you are at high risk for glaucoma
* Heavy alcohol use within the last 6 months (men: more than 4 drinks on any day or more than 14 drinks per week; women: more than 3 drinks on any day or more than 7 drinks per week)
* History of substance use disorder or active use of illicit substances within the last 12 months. Tetrahydrocannabinol (THC)-containing products will not be considered an illicit substance.
* Use of a drug in the monoamine oxidase inhibitor class, currently or within the last 14 days
* Currently pregnant or lactating/breastfeeding; intention to get pregnant in next 24 months; seeking or in active treatment for infertility
* End-stage renal disease on dialysis or CKD class IV or higher (eGFR <30)
* History of valvular heart disease
* Congestive heart failure (any history or current)
* Cirrhosis or symptoms of liver failure in the last 2 years
* Severe pulmonary disease requiring supplemental oxygen
* Quit using nicotine-containing products less than 6 months prior to baseline visit or intention to quit use in the next 2 years
* Use of oral corticosteroids more than 5 days/month in the last 3 months
* Elevated depressive symptoms
* Uncontrolled anxiety symptoms
* Hospitalization for mental illness in the last 24 months
* Diagnosis of dementia or serious mental illness (e.g., schizophrenia, bipolar disorder, severe depression)
* Binge Eating Disorder, Bulimia or Anorexia Nervosa diagnosis or treatment within the last 2 years
* Prior procedure for weight control (including bariatric surgery, devices)
* Use of phentermine, phentermine-containing medication, or anti-obesity medication with similar mechanism of action to phentermine (e.g., phendimetrazine or diethylpropion) in the previous 24 months
* Use of any non-phentermine-containing medications prescribed for weight loss in previous 12 months
* Unstable dose of weight-loss-promoting medications within the last 12 months. Weight-loss-promoting medications are medication prescribed for another condition, but are known to have weight loss effects. Examples would include use of a GLP1 agonist or SGLT2 inhibitor in patients with diabetes; use of topiramate among patients with migraine headaches.
* Use of any stimulant medications in previous 12 months
* Known allergy or intolerance to phentermine or phentermine-containing medication
* Documented or self-reported weight change (gain or loss) of more than 5% of current body weight in the past 3 months
* History of cancer other than non-melanoma skin cancer in the past 5 years
* History of organ transplantation
* Plan to move outside the area in the next two years
* Unable to make changes to diet (e.g., severe food allergies or intolerances; medically necessary aspects of diet incompatible with intervention)
* Already participating in another research study that includes lifestyle changes and/or study medication or has participated in such a study within the last 12 months
* Total body weight that exceeds 400 lbs., precluding use of the digital scale in the lifestyle intervention
* Upper arm circumference that exceeds 50 cm, precluding use of the OMRON HEM 907 XL to measure blood pressure
* Other concern or medical comorbidity that, per discretion of study clinician, would render the participant unfit or unable to safely take part in the 24-month intervention

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in body weight (%) | Baseline to month 24
  The primary outcome for efficacy will be percent weight loss at 24 months of follow-up, relative to body weight (kg) at randomization.
Change in Systolic Blood Pressure (mmHg) | Baseline to month 24
  The primary outcome to address phentermine's impact on a key cardiovascular disease risk factor, blood pressure, will be assessed at 24 months. Staff will measure BP using a standardized protocol with automated BP measurement devices (Omron HEM907XL) and following standard clinical practice guidelines for blood pressure measurement.

SECONDARY OUTCOMES:
Change in resting energy expenditure (REE) / resting metabolic rate (RMR) | Baseline to month 6; Baseline to month 24
  RMR will be measured via indirect calorimetry using the KORR ReeVue (KORR Medical Technologies, Salt Lake City, UT).
Change in cardiac autonomic function | Baseline to month 3; Baseline to month 6; Baseline to month 12; Baseline to month 24
  Change in cardiac autonomic function will be measured using heart rate variability with electrocardiogram (ECG). Heart rate variability (HRV) and resting heart rate (RHR) are noninvasive measures of cardiac autonomic function.
Dependence on study drug (phentermine) | Month 24
  Dependence on study drug will be assessed using the Severity of Dependence Scale (SDS), a brief 5-item validated measure of psychological dependence that has been used for both illegal drugs of abuse and prescription drugs with concern for addiction potential. The score ranges from 0-15 with a higher score denoting a stronger dependence on the study drug.
Change in Systolic Blood Pressure (mmHg) | Baseline to month 6; Baseline to month 12; Baseline to month 18
  To address phentermine's impact on blood pressure over the course of the study, change in systolic blood pressure will be assessed at 6 months using a standardized measurement protocol with automated BP devices and following standard clinical practice guidelines for blood pressure measurement.

OTHER OUTCOMES:
Incident cardiovascular disease or death | Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, Month 21, Month 24
  To address the impact of phentermine on cardiovascular disease and total mortality, participant diagnoses, hospitalizations, treatment, and deaths will be tracked via a combination of self-report and tracking within the electronic medical record.
Change in body weight (%) | Baseline to month 6; Baseline to month 12
  To assess the efficacy of phentermine at intervals throughout the study, percent weight loss at 6 and 12 months of follow-up relative to body weight (kg) at randomization will be measured.
Change in self-reported physical activity levels | Baseline to month 6; Baseline to month 12; Baseline to month 24
  The International Physical Activity (IPAQ) short form is a 7-item index that asks respondents the number of days per week and the amount of time per day spent in vigorous- and moderate-intensity activities and walking, during the seven days prior to the visit. Different levels of physical activity are assigned metabolic equivalent (MET) scores based on the Compendium of Physical Activity and, using MET-minutes, can be converted to both continuous and categorical values

CONTACTS AND LOCATIONS:
Overall Officials: Kristina H Lewis, MD, Principal Investigator — Wake Forest University Health Sciences; Jamy D Ard, MD, Principal Investigator — Wake Forest University Health Sciences; Nicholas M Pajewski, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (4):
- United States (4):
  - Kaiser Permanente Southern California, Los Angeles, California
  - HealthPartners Institute, Saint Louis Park, Minnesota
  - Atrium Health Wake Forest Baptist Weight Management Center, Winston-Salem, North Carolina
  - UT Center for Obesity Medicine and Metabolic Performance, Bellaire, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Young CB, Rives E, Gudzune KA, Jaeger BC, Simmons CG, White BN, Hooker SA, Horn DB, Young DR, Vesely J, Velazquez A, Price C, Cook SD, Martin-Fernandez K, Inzhakova G, Pajewski NM, Ard JD, Lewis KH. The long-term effectiveness of the anti-obesity medication phentermine (LEAP) trial: Rationale, design, and baseline characteristics. Contemp Clin Trials. 2026 Feb;161:108219. doi: 10.1016/j.cct.2026.108219. Epub 2026 Jan 8. PMID 41519431